CLINICAL TRIAL: NCT02345174
Title: An Open Label Positron Emission Tomography (PET) Imaging Study Using 89Zirconium to Investigate the Biodistribution of Anti-HER3 Monoclonal Antibody (mAb) GSK2849330 and Characterize Its Dose-receptor Occupancy Relationship in Subjects With Advanced HER3-Positive Solid Tumors
Brief Title: Immuno Positron Emission Tomography Study of GSK2849330 in Subjects With Human Epidermal Growth Factor Receptor 3-Positive Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 200980
Record Dates: First submitted 2015-01-19; First posted 2015-01-26 (Estimated); Last update posted 2019-02-21 (Actual); Status verified 2019-02

CONDITIONS: Cancer; Neoplasms
Keywords: zirconium; oncology; mAb; receptor occupancy; dose; PET; HER3; 89-Zr; biodistribution; tumours
MeSH Terms: conditions — Neoplasms | interventions — GSK2849330

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Imaging Phase + Continuation Phase (Experimental): In Part 1 of the study, participants will receive a dose of 89Zr-GSK2849330 (Dose 1), with an activity of no more than 37 MegaBequerel (MBq) and a variable total dose of GSK2849330. PET scans will be acquired within 7 days. Two weeks after Dose 1 participants will receive second dose of 89Zr-GSK2849330 (Dose 2) and a variable total dose of GSK2849330. Participants will continue to receive unlabelled GSK2849330 (in Part 2) either at established dose level or as decided by medical monitor.
  Interventions: Drug: GSK2849330; Drug: 89Zr-GSK2849330

INTERVENTIONS:
Drug: GSK2849330 — GSK2849330 solution (100 mg/mL) for infusion diluted in 0.9% sodium chloride to the appropriate concentration for the dose.
Drug: 89Zr-GSK2849330 — 89Zr-GSK2849330 solution for intravenous administration diluted with GSK2849330 Solution for Infusion (unlabelled GSK2849330) with a target radioactivity of 37MBq and a total antibody concentration of 0.4 mg/mL or 1.2 mg/mL.

SUMMARY:
Human epidermal growth factor receptor 3 (HER3) expression is seen across a wide variety of solid malignancies and is associated with poor prognosis. Up-regulation of HER3 expression and activity is also associated with resistance to multiple pathway inhibitors. GSK2849330, a monoclonal antibody (mAb) targeting HER3, is a new agent for subjects whose tumors express HER3. This study aims to characterise the biodistribution and dose-receptor occupancy relationship of GSK2849330 in patients with advanced HER3 expressing solid tumours via the use of PET imaging. This study will be conducted in two parts. Part 1 will be the imaging phase where each subject will receive two doses of GSK2849330 containing both Zirconium-89 (89Zr) labelled GSK2849330 and unlabeled GSK2849330. The amount of unlabeled GSK2849330 present in each dose will be varied to explore the effect on target mediated uptake of 89Zr into HER3 expressing tissues and tumors. Subjects will then proceed to the continuation phase (Part 2) for continued treatment with unlabelled GSK2849330. The study is planned to enroll approximately 12-15 subjects.

ELIGIBILITY:
Inclusion Criteria

* Males and females >=18 years of age (at the time consent is obtained).
* Written informed consent provided.
* Performance Status score of 0 or 1 according to the Eastern Cooperative Oncology Group (ECOG) scale.
* Sufficient archival tumor specimen is available for HER3 immunohistochemistry (IHC) analysis, or subject is willing to undergo a tumor biopsy for HER3 IHC analysis.
* Subjects must have tumours with documented HER3 expression on the cell surface (1+, 2+ or 3+) of the invasive component of tumour (either on archival tissue or a fresh biopsy) using an analytically validated IHC assay by central laboratory.
* Histologically or cytologically confirmed diagnosis of solid tumour malignancy for which no standard therapeutic alternatives exist.
* Adequate baseline organ functions
* Left ventricular ejection fraction (LVEF) >=50% by Echocardiogram (ECHO) or Multi gated acquisition scan (MUGA).
* Subjects must have at least two measurable lesions on Computed tomography (CT) or Magnetic resonance imaging (MRI) scan with a shortest axis of at least 20 millimeter (mm).

Exclusion Criteria:

* Subjects with leptomeningeal or brain metastases or spinal cord compression
* Prior HER3- directed treatment (HER2- or EGFR-directed treatment is acceptable).
* Unresolved toxicity greater than National Cancer Institute - Common Terminology Criteria for Adverse Events (NCI-CTCAE), version 4.0 Grade 1 from previous anti-cancer therapy
* Known or suspected hypersensitivity reaction to prior biologic therapy
* Evidence of another active malignancy (excludes non-melanoma skin cancer).
* Concurrent medical condition that would jeopardize compliance with the protocol.
* Receiving concurrent anti-tumor therapies, or chronic immunosuppressive therapies (includes daily steroid doses in excess of 20 milligram (mg)/day of prednisolone).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2015-03-19 (Actual); Primary Completion 2016-06-02 (Actual); Study Completion 2016-06-02 (Actual)

PRIMARY OUTCOMES:
Standardized Uptake Value (SUV). | Up to Day 21
  Regions of interest (RoI) will be outlined from PET-CT images to represent the tissue radioactivity concentration through the values of SUVmean and SUVpeak.
Volume of region of interest. | Up to Day 21
  RoIs will be outlined to represent whole organs and include the volumes encircled

SECONDARY OUTCOMES:
Anatomical localization of radiolabel. | Up to Day 21
  Anatomical localization of radiolabel will be evaluated to establish dose-dependency of inhibition of target mediated uptake of 89Zr-GSK2849330 by unlabeled GSK2849330.
Uptake of-GSK2849330 in tumors using pharmacometric model | Up to Day 21
  Uptake of GSK2849330 in tumors will be estimated to establish dose-dependency of inhibition of target mediated uptake of 89Zr-GSK2849330 by unlabeled GSK2849330.
Change in uptake parameters in response to the dose difference between dose 1 and 2. | Up to Day 21
  Change in uptake parameters following dose 1 and 2 will estimated to establish dose-dependency of inhibition of target mediated uptake of 89Zr-GSK2849330 by unlabeled GSK2849330.
Average radioactivity concentration in whole blood and plasma | Up to Day 21
  Average radioactivity concentration will be determined and expressed as SUV and is equal to tissue radioactivity concentration normalized by administered amount of radioactivity per body weight.
Tumor features assessment | Up to Day 21
  Features of tumor will include central necrosis, irregular shape, non-uniform uptake and lesion ID
Composite of pharmacokinetic (PK) parameters of GSK2849330 | Predose, and at 1, 3, 6, 12 and 24 hours post dose.
  Measurements will include: maximum observed plasma concentration (Cmax), time to Cmax (tmax), area under the plasma concentration-time curve (AUC(0-t), AUC(0-Tau) (repeat dosing) and/or AUC(0-Infinity) (single dose), apparent terminal phase elimination rate constant (lambda z) and apparent terminal phase half-life (t½)
Organ dose measured in milliSievert (mSv) for each organ | Up to Day 21
Effective dose value measured in mSv | Up to Day 21
Overall incidence of Adverse events (AEs) and Serious Adverse events (SAEs) | Average of 6 months
  AEs and SAEs will be collected from the time the first dose of study treatment is administered until 45 days following discontinuation of study treatment
Change from baseline in laboratory parameters | Baseline and up to 6 months
  Clinical laboratory tests will include clinical chemistry, routine urinalysis, haematology laboratory evaluations and additional parameters
Left ventricular ejection fraction (LVEF) assessment | Average of 6 months
  LVEF will be assessed as a measure of safety and tolerability measured by echocardiography (ECHO) or multi gated acquisition (MUGA) scans
Vital signs monitoring. | Average of 6 months
  Vital sign measurements will include systolic and diastolic blood pressure (BP), temperature, and pulse rate
Serum titer of the anti-GSK2849330 antibodies. | Average of 6 months
  Samples will be analyzed for the presence of anti-GSK2849330 antibodies using a validated immunoelectrochemiluminescent (ECL) assay.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline; GSK Clinical Trials, Study Director — GlaxoSmithKline (for GlaxoSmithKline; Human Genome Sciences Inc., a GSK Company; Sirtris, a GSK Company; Stiefel, a GSK Company; ViiV Healthcare)
Locations (1):
- GSK Investigational Site, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com

REFERENCES:
- [Background] Menke-van der Houven van Oordt CW, McGeoch A, Bergstrom M, McSherry I, Smith DA, Cleveland M, Al-Azzam W, Chen L, Verheul H, Hoekstra OS, Vugts DJ, Freedman I, Huisman M, Matheny C, van Dongen G, Zhang S. Immuno-PET Imaging to Assess Target Engagement: Experience from 89Zr-Anti-HER3 mAb (GSK2849330) in Patients with Solid Tumors. J Nucl Med. 2019 Jul;60(7):902-909. doi: 10.2967/jnumed.118.214726. Epub 2019 Feb 7. PMID 30733323
- See also: Results for study 200980 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/200980?search=study&b'study_ids=200980'#rs